CLINICAL TRIAL: NCT01893021
Title: Family Planning Knowledge, Attitudes, and Practices of HIV+ and HIV- Postpartum Malawian Women
Brief Title: Family Planning Knowledge, Attitudes, and Practices of Postpartum Malawian Women
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Jennifer Tang, MD, MSCR, Research Assistant Professor, University of North Carolina, Chapel Hill
Other Study IDs: 13-1084; 1R25TW009340-01 (NIH); P30AI050410 (NIH)
Record Dates: First submitted 2013-06-26; First posted 2013-07-08 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postpartum Malawian women

SUMMARY:
The purpose of this study is to understand the family planning needs and practices of postpartum Malawian women, with a focus on long-acting reversible contraception (LARC).

Hypotheses:

1. Postpartum women who are older, who have a history of unintended pregnancy, who do not desire another child within 2 years, and who were counseled about LARC during their pregnancy are more likely to have interest in using LARC.
2. Postpartum women who are older are more likely to be aware of LARC methods.
3. HIV+ postpartum Malawian women will have similar knowledge about LARC as postpartum Malawian women who are HIV-.

DETAILED DESCRIPTION:
This study is a prospective cohort study of 630 postpartum Malawian women. Since our focus is on HIV+ women, HIV+ participants will be recruited in a 1:2 ratio, with a total of 210 HIV+ women and 420 HIV- women. We will recruit in the postpartum ward of Bwaila Maternity Hospital in Lilongwe, Malawi. Participants will complete a baseline survey about demographics, reproductive health history, and family planning knowledge, attitudes, and practices. At 3, 6, and 12 months postpartum, we will complete follow-up phone calls to determine what family planning methods they are using and if they encountered any barriers to receiving LARC if they had been interested in using them.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to the postpartum ward at Bwaila Maternity Hospital
2. Live birth ≥28 weeks gestational age within past 4 weeks
3. Fluent in English or Chichewa
4. Age 18-45 years
5. Access to a working phone number
6. Willingness to be contacted by phone for up to one year postpartum

Exclusion Criteria:

1. History of female sterilization via tubal ligation or hysterectomy
2. Prisoner
3. History of mental disability
4. Serious illness that would prevent participation in the opinion of the Principal Investigator

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Our study population will be a sample of 210 HIV+ and 420 HIV- postpartum Malawian women.
Sampling Method: Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Knowledge about the intrauterine device (IUD) and contraceptive implant | Upon enrollment
  A 14-question test about the IUD and implant will be administered to all study participants upon enrollment.

SECONDARY OUTCOMES:
Proportion of women using intrauterine device (IUD) and contraceptive implant | 3, 6, and 12 months postpartum
  We will compare the proportions of HIV+ and HIV- women who are using the IUD and implant at 3, 6, and 12 months postpartum.
Barriers to receiving intrauterine device (IUD) and contraceptive implant | Up to 12 months postpartum
  Descriptive statistics will be used to analyze the reasons given for not receiving the IUD or implant at 3, 5, and 12 months postpartum if a woman had wanted to use it.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tang, MD, MSCR, Principal Investigator — University of North Carolina, Chapel Hill; Mina Hosseinipour, MD, MPH, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- Bwaila Maternity Hospital, Lilongwe, Malawi

REFERENCES:
- [Derived] Tang JH, Kopp DM, Stuart GS, O'Shea M, Stanley CC, Hosseinipour MC, Miller WC, Mwale M, Kaliti S, Bonongwe P, Rosenberg NE. Association between contraceptive implant knowledge and intent with implant uptake among postpartum Malawian women: a prospective cohort study. Contracept Reprod Med. 2016 Aug 10;1:13. doi: 10.1186/s40834-016-0026-1. eCollection 2016. PMID 29201402